CLINICAL TRIAL: NCT00930293
Title: Personalizing Treatment of Depression Complicated by Panic Features-Pilot Study
Brief Title: Efficacy and Feasibility of a Personalized Treatment for Depression With Co-Occurring Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jill Cyranowski, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH085874 (NIH); R01MH085874 (NIH); MH085874-01; PRO08070009; PCC: DSIR 84-CT
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Depression; Anxiety
Keywords: Interpersonal Psychotherapy
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Interpersonal Psychotherapy; Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personalized Depression Care (Experimental): Participants will receive interpersonal psychotherapy for depression with panic and anxiety symptoms (IPT-PS) and standard antidepressant medication (citalopram) treatment.
  Interventions: Behavioral: Interpersonal Psychotherapy for Depression with Panic and Anxiety Symptoms (IPT-PS); Drug: Citalopram hydrobromide
- Standard Depression Care (Active Comparator): Participants will receive brief supportive psychotherapy (BSP) and standard antidepressant medication (citalopram) treatment.
  Interventions: Behavioral: Brief Supportive Psychotherapy (BSP); Drug: Citalopram hydrobromide

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for Depression with Panic and Anxiety Symptoms (IPT-PS) — 16 weekly IPT-PS sessions, each lasting approximately 45 minutes
  Arms: Personalized Depression Care
Behavioral: Brief Supportive Psychotherapy (BSP) — 16 weekly BPS sessions, each lasting approximately 45 minutes
  Arms: Standard Depression Care
Drug: Citalopram hydrobromide — A 20-week regimen of citalopram hydrobromide monotherapy on a flexible dosing schedule ranging from 10 to 60 mg/day
  Other Names: Celexa

SUMMARY:
This study will examine the feasibility and efficacy of a personalized psychotherapy treatment for people with depression and co-occurring anxiety.

DETAILED DESCRIPTION:
Approximately one half of all depressed psychiatric patients also meet the criteria for an anxiety disorder. Compared to people with only depression, people with both depression and panic features experience poorer psychological and social functioning, a greater risk of suicide, less response to medication and therapy treatment, and a greater risk of recurring symptoms. Because people with depression and co-occurring anxiety features do not achieve full symptom remission with either medication or therapy alone, this study will use a treatment that combines the two. A commonly used type of depression medication called a selective serotonin reuptake inhibitor (SSRI) will be combined with a specialized therapy developed to address depression with co-occurring symptoms of panic, anxiety, and avoidance. This study will also test a computer-based method of assessing mood and anxiety symptom profiles and outcomes to determine whether participants find this method acceptable and clinicians find it useful.

Participation in this study will last 20 weeks, with follow-up visits occurring 4 and 8 months after starting. Participants will be randomly assigned to receive either an individualized therapy for depression and anxiety, called interpersonal psychotherapy for depression with panic and anxiety symptoms (IPT-PS), or a standard therapy for depression, called brief supportive psychotherapy (BSP). All participants will complete up to 16 therapy sessions and receive a standard SSRI treatment with the medication citalopram hydrobromide. During the IPT-PS treatment, a study therapist will examine regular computer updates of depression and anxiety scores for participants and talk to them about identifying and addressing life stressors that trigger symptoms. During the BSP treatment, a study therapist will encourage participants to arrive at their own solutions by emphasizing the participants' strengths and examining what has worked in the past.

Participants will complete assessments weekly during the 20 weeks of the study intervention and at 4- and 8-month follow-up visits. These assessments will include self-report questionnaires about symptoms, medication side effects, and treatment adherence; vital sign and weight measurements; and a clinical interview. Regular assessments of medication effectiveness and side effects will occur every 1 to 4 weeks. Starting at the second study visit, participants will also complete monthly computer-based questionnaires about depression and anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Currently in an episode of nonpsychotic major depression, as defined by the DSM-IV and documented by both the Structured Clinical Interview for Axis I, DSM-IV Disorders (SCID) and by a rating of greater than 15 on the 25-item Hamilton Rating Scale for Depression (HRSD)
* Panic spectrum risk category of at least 7, as defined by the Panic-Agoraphobic Spectrum Self-Report (PAS-SR), last month version
* Not currently receiving effective treatment
* Participants with suicidal ideation are eligible as long as outpatient treatment is deemed safe.

Exclusion Criteria:

* History of manic or hypomanic episode(s)
* History of schizophrenia or schizoaffective disorder
* Mood disorder due to a general medical condition or induced by substance use
* Presence of psychosis
* Current pregnancy or plans to become pregnant
* Current primary diagnosis of anorexia nervosa or bulimia nervosa (this does not include an eating disorder not otherwise specified [NOS])
* Current primary diagnosis of severe obsessive-compulsive disorder (OCD), as determined by clinician evaluation of symptom severity and temporal onset of symptoms
* Drug or alcohol abuse or dependence within the past 3 months (participants with episodic abuse related to mood episodes will not be excluded)
* Satisfies full DSM-IV criteria for antisocial personality disorder, as determined by SCID-II evaluation
* Requires inpatient treatment because of suicidal risk or psychotic symptoms (current suicidal thinking or parasuicidal behavior is not exclusionary if, in clinician judgment, it can be managed on an outpatient basis)
* Any of the following medical conditions:

  1. An index episode that is secondary to the effect of medically prescribed drugs, i.e., reserpine, antihistamines, etc.
  2. Presence of significant uncontrolled medical illness including cardiovascular disorder, kidney or liver disease, epilepsy, untreated hypertension, or unstabilized endocrine disease (stable medical conditions such as well-controlled diabetes or HIV positive status are not exclusionary provided the participant meets other inclusion and exclusion criteria)
  3. Current treatment with a pharmacologic, over-the-counter, or herbal therapy for depression or anxiety (unless the participant wishes to discontinue an ineffective treatment)
* History of poor or failed treatment response to an adequate dose and duration of citalopram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M. Cyranowski, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Personalized Depression Care: Participants will receive interpersonal psychotherapy for depression with panic and anxiety symptoms (IPT-PS) and standard antidepressant medication treatment.
  Interpersonal Psychotherapy for Depression with Panic and Anxiety Symptoms (IPT-PS): 16 weekly IPT-PS sessions, each lasting approximately 45 minutes
  Citalopram hydrobromide: A 20-week regimen of citalopram hydrobromide monotherapy on a flexible dosing schedule ranging from 10 to 60 mg/day
- Standard Depression Care: Participants will receive brief supportive psychotherapy (BSP) and standard antidepressant medication treatment.
  Brief Supportive Psychotherapy (BSP): 16 weekly BPS sessions, each lasting approximately 45 minutes
  Citalopram hydrobromide: A 20-week regimen of citalopram hydrobromide monotherapy on a flexible dosing schedule ranging from 10 to 60 mg/day
Period: Overall Study
Arm/Group | Personalized Depression Care | Standard Depression Care
Started | 24 | 26
Completed | 17 | 19
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Depression Care | Standard Depression Care | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.37 (11.41) | 31.09 (10.27) | 30.74 (10.72)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 5 | 8 | 13
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Meeting Depression Remission Criteria
Description: Depression remission defined as 3 consecutive weeks of HRSD-17 scores that on average, < or = 7
Time Frame: Measured at baseline and weekly for up to 20 weeks of acute treatment
Measure: Number; unit: participants
Arm/Group | Personalized Depression Care | Standard Depression Care
Number analyzed (Participants) | 24 | 26
participants | 10 | 15

2. Secondary Outcome: Weeks to Depression Remission
Description: Kaplan-Meier survival analyses to determine time to depression remission (defined as average HRSD-17 score < or = 7 for three consecutive weeks).
  Analyses run with the full intent to treat sample (censoring patients who dropped out at time of termination)
Time Frame: Measured at baseline and weekly for up to 20 weeks of treatment
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Personalized Depression Care | Standard Depression Care
Number analyzed (Participants) | 24 | 26
weeks | 13.99 (1.47) | 11.59 (1.31)

ADVERSE EVENTS:
Arm/Group | Personalized Depression Care | Standard Depression Care
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 1/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personalized Depression Care (N=24) | Standard Depression Care (N=26)
Unexplained Visual Disturbance (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes